CLINICAL TRIAL: NCT03436979
Title: The NeuGuide™ System for Vaginal Colpopexy in the Treatment of Uterine Prolapse Post-Market Surveillance Clinical Study
Brief Title: The NeuGuide™ System for Vaginal Colpopexy in the Treatment of Uterine Prolapse
Status: Completed | Type: Observational
Sponsor: Pop Medical Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: 06-CLP-0098
Record Dates: First submitted 2018-01-23; First posted 2018-02-19 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Uterine Prolapse Without Vaginal Wall Prolapse
Keywords: prolapse; sacrospinous fixation; minimally invasive
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Subjects: Subjects who are undergoing surgical treatment for uterine prolapse will be included in the study and will be treated using the NeuGuide™ System.
  Interventions: Device: NeuGuide™ System

INTERVENTIONS:
Device: NeuGuide™ System — The NeuGuide™ device is indicated for anchoring sutures to ligaments of the pelvic floor.
  Other Names: transvaginal sacrospinous ligament fixation

SUMMARY:
The objective of the study is to assess the long term safety, durability of clinical effectiveness and cost effectiveness of the NeuGuide™ system when used for vaginal colpopexy in the treatment of uterine prolapse.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with POP-Q C point greater than (-) 1 cm.
2. Patients who have previously had a partial hysterectomy in which the cervix is intact may be included in this study.
3. Non-pregnant female (female of child bearing potential must have a negative pregnancy test).
4. Patient understands the nature and potential hazards of the procedure and provides written informed consent prior to any study specific assessments.
5. Patient is able to complete written questionnaires.
6. Patient is willing and able to comply with the specified study requirements and follow-up assessments, and can be contacted by telephone.

Exclusion Criteria:

1. Known diagnosis of reproductive tract abnormalities.
2. Prior pelvic radiation therapy, any malignancy or active pelvic inflammatory disease.
3. Known history of severe Pelvic Inflammatory Disease (PID).
4. Prior total hysterectomy.
5. Prior pelvic prolapse surgery using synthetic mesh.
6. Pathological PAP in the past year.
7. Moderate or severe bacterial cervicitis.
8. Moderate or severe pelvic pain (> 3 on VAS).
9. Severe morbid obesity (BMI >45).
10. Temperature > 38°C (oral or equivalent), sepsis, or active infection requiring IV anti-microbial treatment.
11. Significant cognitive impairment.
12. Active malignancy other than non-melanoma skin cancer.
13. Planned surgery (more than a minor one) in the next 30 days.
14. Patient has a known hypersensitivity to device materials (Nickel, suture material).
15. Moribund patient or patient with severe or deteriorating damage in critical body systems.
16. Any condition that in the judgment of the investigators would interfere with the subject's ability to provide informed consent, comply with study instructions, place the subject at increased risk, or which might confound interpretation of study results.
17. Concurrent enrollment in another device or drug trial that has not completed the primary endpoint or clinically interferes with the current study endpoints.

Ages: 36 Years to 84 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Must have uterine prolapse
Study Population: Subjects who are undergoing surgical treatment for uterine prolapse.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
A composite of the Pelvic Organ Prolapse Quantification (POP-Q) C point score, patient-rated symptom of vaginal bulging after vaginal colpopexy performed using the NeuGuide™ and the absence of further surgical therapy for uterine prolapse. | 12 months
  Primary composite performance outcome
The number of device / procedure related Serious Adverse Events (SAE). | 30 days
  Primary safety of surgical implantation as reflected by adverse events
The number of Serious Adverse Events and Adverse Events. | 12 months
  Primary safety of NeuGuide treatment as reflected by adverse events

SECONDARY OUTCOMES:
Change in mean POP-Q C point score from baseline (cm). | one month
  Secondary anatomical performance of the NeuGuide treatment
Change in mean POP-Q C point score from baseline (cm). | 6 months
  Secondary anatomical performance of the NeuGuide treatment
Change in mean POP-Q C point score from baseline (cm). | 12 months
  Secondary anatomical of the NeuGuide treatment
Change in mean POP-Q C point score from baseline (cm). | 24 months
  Secondary anatomical performance of the NeuGuide treatment outcome
Change in mean POP-Q C point score from baseline (cm). | 36 months
  Secondary anatomical performance of the NeuGuide treatment
Number of subjects who require surgical therapy of uterine prolapse or urinary incontinence. | 36 months
  Secondary performance: durability of the NeuGuide treatment
Number of subjects in whom the primary symptomatic reason for repair of prolapse persists. | 12 months
  Secondary symptomatic performance of the NeuGuide treatment
The time utilization of staff performing the NeuGuide procedure. | one month
  Secondary outcome: Cost performance of the procedure
The POP-Q Stage Score calculated from POP-Q measurements, where the Stages of POP-Q system measurement are as follows: Stage 0 no prolapse is demonstrated Stage 1 the most distal portion of the prolapse is more than 1 cm above the level of the hymen | Baseline
  Secondary outcome: POP-Q Stage Score.
The POP-Q Stage Score calculated from POP-Q measurements, where the Stages of POP-Q system measurement are as follows: Stage 0 no prolapse is demonstrated Stage 1 the most distal portion of the prolapse is more than 1 cm above the level of the hymen | one month
  Secondary outcome: POP-Q Stage Score.
The POP-Q Stage Score calculated from POP-Q measurements, where the Stages of POP-Q system measurement are as follows: Stage 0 no prolapse is demonstrated Stage 1 the most distal portion of the prolapse is more than 1 cm above the level of the hymen | 12 months
  Secondary outcome: POP-Q Stage Score.
The POP-Q Stage Score calculated from POP-Q measurements, where the Stages of POP-Q system measurement are as follows: Stage 0 no prolapse is demonstrated Stage 1 the most distal portion of the prolapse is more than 1 cm above the level of the hymen | 24 months
  Secondary outcome: POP-Q Stage Score.
The POP-Q Stage Score calculated from POP-Q measurements, where the Stages of POP-Q system measurement are as follows: Stage 0 no prolapse is demonstrated Stage 1 the most distal portion of the prolapse is more than 1 cm above the level of the hymen | 36 months
  Secondary outcome: POP-Q Stage Score.

CONTACTS AND LOCATIONS:
Overall Officials: James C Leiter, M.D., Study Director — Avania
Locations (15):
- United States (11):
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Mount Auburn Hospital, Cambridge, Massachusetts
  - Maimonides Medical Center, Brooklyn, New York
  - South Nassau Community Hospital Cancer Center, Valley Stream, New York
  - Cleveland Clinic Cleveland, Cleveland, Ohio
  - The Institute for Female Pelvic Medicine and Reconstructive Surgery, Allentown, Pennsylvania
  - Female Pelvic Health Center, Newtown, Pennsylvania
  - Walnut Hill OB/GYN Associates, Dallas, Texas
  - INOVA Women's Hospital, Falls Church, Virginia
- Germany (3):
  - Krankenhaus Waldfriede, Berlin-Zehlendorf
  - Isar Kliniken GmbH, München
  - St. Joseph Krankenhaus, Tempelhof
- Soroka Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data a available to other researchers.